CLINICAL TRIAL: NCT03834376
Title: Pimodivir (JNJ-63623872) Pre Approval Access_Single Patient Access (SPR) for Patients Diagnosed With H7N9 Influenza A Infection
Brief Title: Pre-Approval Access to Pimodivir for the Treatment of Patients With H7N9 Influenza A Infection
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108461; 63623872FLZ4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: H7N9 Subtype of Influenza A Virus
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Pimodivir — Pimodivir will be administered as tablets taken orally, twice daily (2 tablets of 300 milligram [mg]) over a time period of 5 days.
  Other Names: JNJ-63623872

SUMMARY:
The purpose of this program is to provide pre-approval access to pimodivir for the treatment of a patient(s) with H7N9 influenza A infection. Pre-approval access pertains to provision for therapeutic use of an investigational product prior to its marketing authorization. Such access may be considered for eligible patients with serious/life-threatening diseases or conditions, where alternative treatments do not exist or have been exhausted.

ELIGIBILITY:
Inclusion Criteria:

* The patient has an H7N9 Influenza A infection
* The patient has no known severe hepatic impairment

Exclusion Criteria:

- Any other Influenza A sub-strains other than H7N9

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult